CLINICAL TRIAL: NCT03194919
Title: The Effect of Negotiating a Quit Date on Attempting to Quit Smoking
Brief Title: Negotiating a Quit Date or Not in Online Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Håvar Brendryen, Senior Research Scientist, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFR 228158/H10-B
Record Dates: First submitted 2017-06-19; First posted 2017-06-21 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Nicotine Dependence, Cigarettes
Keywords: online intervention; e-Health; negotiating quit date
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants receive one out of two versions of a web-based smoking cessation program. Either with or without the option of negotiating and re-negotiating the quit date.
Masking Description: The recruitment procedure and the treatment is fully automated and delivered by web, e-mail and SMS-textmessages - i.e., the participant is not contacted by any care providers, investigators or assessors during recruitment or treatment
  - and data are collected by means of web-based questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negotiating quit date (Experimental): Endre: a digital smoking cessation counsellor
  Interventions: Other: Endre: a digital smoking cessation counsellor
- Preset quit date (Active Comparator): Endre: a digital smoking cessation counsellor
  Interventions: Other: Endre: a digital smoking cessation counsellor

INTERVENTIONS:
Other: Endre: a digital smoking cessation counsellor — A comprehensive 25-session intervention delivered by web, e-mail and SMS-text messages. Sessions are released one each day for 18 days, and then every second day for 14 days. Intervention content is tailored based on user input and individual usage pattern. The intervention is described in detail in Holter, Johansen & Brendryen (2016). How a fully automated eHealth program simulates three therapeutic processes: A case study. Journal of Medical Internet Research 18 (6).

SUMMARY:
The primary purpose of the current study is to test the effect of providing users of automated web-based smoking cessation interventions with the option of negotiating and re-negotiating the quit date.

DETAILED DESCRIPTION:
Web- and mobile phone health behavior change interventions, including smoking cessation programs, offer great promise, but little is known about how such interventions should be designed to increase their efficacy

The primary purpose of the current study is to test the effect of providing users of automated web-based smoking cessation interventions with the option of negotiating and re-negotiating the quit date.

The investigators propose a 2-arm RCT with 1500 adult study participants that all receive a best practices web-based smoking cessation program designed for use on smart phones (web-app). The intervention includes a ten day/session preparation phase (participants continue smoking) as well as a four week post-cessation follow-up phase (14 sessions). The post-cessation phase will only be given to participants that report an initial quit attempt. Participants will be randomized to two versions of the intervention: 1) A version that does not provide participants with the option of negotiating the quit day (the preparation phase is fixed to ten days/sessions); or 2) a version that provides the participants with the option of negotiating/re-negotiate the quit day on three occasions. The three occasions are on the first day/session of the intervention, on the fourth day/session of the intervention and on the eleventh day/session of the intervention. The primary outcome is making a quit attempt.

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* being a current smoker
* determined to or considering to quit smoking
* provide valid e-mail address
* provide valid norwegian cell phone number
* complete a baseline questionnaire
* start using the intervention (pushing the next page button one time or more on the first session provided

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Quit attempt | Within 6 weeks after starting the first session of the intervention
  User report a quit attempt

SECONDARY OUTCOMES:
Number of sessions in preparation phase completed | Within 6 weeks after starting the first session of the intervention
  Ten sessions are available
Number of sessions in preparation phase started | Within 6 weeks after starting the first session of the intervention
  Ten sessions are available

CONTACTS AND LOCATIONS:
Overall Officials: Håvar Brendryen, PhD, Principal Investigator — University of Oslo
Locations (2):
- Department of Addictology, 1st Faculty of Medicine, Charles University, Prague, Czechia
- The Norwegian Centre for Addiction Research, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holter MT, Johansen A, Brendryen H. How a Fully Automated eHealth Program Simulates Three Therapeutic Processes: A Case Study. J Med Internet Res. 2016 Jun 28;18(6):e176. doi: 10.2196/jmir.5415. PMID 27354373
- See also: Official home page for PI at host institution — https://www.sv.uio.no/psi/english/people/aca/haavabre/index.html